CLINICAL TRIAL: NCT05114512
Title: Rural Access to Physical Therapy for Osteoarthritis Rehabilitation
Brief Title: Rural Access to Physical Therapy for Osteoarthritis Rehabilitation - Pilot
Acronym: RAPTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Pittsburgh Medical Center Rehabilitation Institute (Unknown)
Responsible Party: Principal Investigator, Allyn Bove, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY21050074
Record Dates: First submitted 2021-09-29; First posted 2021-11-10 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis, Knee
Keywords: arthritis; physical therapy; rehabilitation; rural; telehealth; telerehabilitation; knee; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Single cohort of 27 individuals
Masking Description: This is a single-group study; therefore, no masking is possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RAPTOR Physical Therapy Intervention (Experimental): RAPTOR intervention: hybrid in-person + telehealth physical therapy care for rural-dwelling individuals with knee osteoarthritis
  Interventions: Other: RAPTOR protocol: hybrid in-person + telehealth physical therapy services

INTERVENTIONS:
Other: RAPTOR protocol: hybrid in-person + telehealth physical therapy services — All participants will receive the RAPTOR intervention, which includes 2 in-person physical therapy visits and 8 telerehabilitation visits. Participants will attend an initial in-person PT evaluation to meet their provider, receive a hands-on assessment of their impairments and functional limitations, and receive instruction in an initial home exercise program. The remainder of their visits will be completed remotely, using a telerehabilitation platform. At the conclusion of care, the patient will return to the clinic for a follow-up assessment and training on their final home exercise program.

SUMMARY:
This is a pilot study involving a hybrid in-person + telerehabilitation intervention for rural adults with knee osteoarthritis. The primary purpose is to demonstrate feasibility and safety of the RAPTOR program, and the secondary purpose is to estimate clinical effectiveness of the RAPTOR program on participants' pain, function, and quality of life.

DETAILED DESCRIPTION:
The purpose of the RAPTOR pilot study is to determine feasibility of a rural telerehabilitation intervention by assessing (1) attendance rate for telerehabilitation visits among participants in the pilot program; (2) participants satisfaction with the program; and (3) participant outcomes regarding pain, function, and quality of life. This pilot study will provide preliminary data to support efforts to obtain external funding for a future randomized trial comparing traditional physical therapy (PT) to the RAPTOR approach.

The primary purpose of the RAPTOR pilot study is to demonstrate feasibility and safety of the RAPTOR program in rural adults with knee osteoarthritis (KOA). The secondary purpose is to estimate clinical effectiveness of the RAPTOR program on participants' pain, function, and health-related quality of life. This will enable the investigators to determine a sample size estimate for a future trial comparing RAPTOR to a traditional face-to-face physical therapy approach in this population.

Specific Aim 1: To assess feasibility of the Rural Access to Physical Therapy for Osteoarthritis Rehabilitation (RAPTOR) program in delivering a hybrid telerehabilitation program to rural people with KOA.

Hypothesis 1: Participants in the RAPTOR program will attend at least 80% of study-related in-person and telerehabilitation visits, and will experience no serious adverse events.

Specific Aim 2: To determine preliminary clinical effectiveness of the RAPTOR program by assessing pain, physical function, and health-related quality of life via patient-reported and performance-based outcomes.

Hypothesis 2: A majority of RAPTOR participants will demonstrate clinically meaningful improvement in patient-reported pain, physical function, and/or health-related quality of life.

ELIGIBILITY:
Potential participants who meet all of the following criteria will be included:

* Participant meets American College of Rheumatology criteria for the clinical diagnosis of knee osteoarthritis
* Participant's home address is in a rural (non-core) western Pennsylvania county
* Participant is willing to travel to Centers for Rehab Services - Bedford clinic for two face-to-face sessions with a licensed physical therapist
* Participant has access to high-speed internet and/or LTE wireless service and a device (tablet, computer, or smartphone) to access the telerehabilitation platform
* Participant is aged 40 or over

Potential participants will be excluded if any of the following criteria apply:

* Chronic neurological disorder affecting balance or coordination
* Any other disorder that affects balance or gait
* Two or more falls in the past 12 months, OR sought medical attention for any fall within the past 12 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Recruitment Target | Through study completion, which is anticipated to take approximately 1 year.
  The investigators' recruitment target is 27 participants, and this outcome will be successful upon enrollment of the 27th participant. This outcome will be used as one component of the overall summary outcome of "feasibility", which is defined as success in all 5 primary outcomes.
Visit Attendance (75% or higher) | Through study completion, which is anticipated to take approximately 1 year.
  The percentage of physical therapy visits attended, divided by the number of scheduled visits (10) for each participant. This outcome will be successful if mean visit attendance among all participants is at least 75%. This outcome will be used as one component of the overall summary outcome of "feasibility", which is defined as success in all 5 primary outcomes.
Telehealth Usability Questionnaire | Measured at post-treatment (last visit, approximately 10 weeks after enrollment)
  The Telehealth Usability Questionnaire (5/7) is a self-reported questionnaire used to assess participant satisfaction with the telehealth services received. It contains 21 items, each rated on a 7-point scale ranging from "strongly disagree" (1 point) to "strongly agree" (7 points). The items are summed to create a total score ranging from 7 - 147 points, with higher numbers indicating greater usability of the telehealth services. This outcome will be successful if the average item rating across all participants is at least 5/7. This outcome will be used as one component of the overall summary outcome of "feasibility", which is defined as success in all 5 primary outcomes.
Study-Related Adverse Events / Serious Adverse Events | Through study completion, which is anticipated to take approximately 1 year.
  This outcome will be successful if there are zero study-related adverse events and serious adverse events among the 27 participants. This outcome will be used as one component of the overall summary outcome of "feasibility", which is defined as success in all 5 primary outcomes.
Clinically Important Improvement on ONE Functional Outcome Measure | Baseline (measured at first visit) and post-treatment (measured at last visit, approximately 10 weeks later)
  The final component of the overall primary outcome of feasibility will be met if each participant achieves mean improvement on at least one functional outcome measure that exceeds the minimum clinically important difference. This may occur on a self-reported outcome measure (the KOOS, described below) or a performance-based outcome measure (30-second chair stand test, timed stair climb test, Timed Up and Go test, 40-meter fast-paced walk test, 6-minute walk test). All of these outcome measures are individually considered to be Secondary Outcome Measures and are described below in greater detail.

SECONDARY OUTCOMES:
Functional outcome measure: 30-second chair stand test | Baseline (measured at first visit) and post-treatment (measured at last visit, approximately 10 weeks later)
  Measures the number of times the participant can stand up and sit down from a chair in a 30-second period.
Functional outcome measure: Timed stair climb test | Baseline (measured at first visit) and post-treatment (measured at last visit, approximately 10 weeks later)
  Measures the number of seconds it takes the participant to climb and descend 1 full flight of standard stairs.
Functional outcome measure: Timed Up and Go (TUG) | Baseline (measured at first visit) and post-treatment (measured at last visit, approximately 10 weeks later)
  Measures the number of seconds it takes for the participant to stand up from a chair, walk 3 meters, turn around, walk 3 meters back to the chair, and sit back down in the chair.
Functional outcome measure: 40-meter fast-paced walk test | Baseline (measured at first visit) and post-treatment (measured at last visit, approximately 10 weeks later)
  Measures the number of seconds it takes the participant to walk 40 meters at what the participant considers to be a "fast pace".
Functional outcome measure: 6-minute walk | Baseline (measured at first visit) and post-treatment (measured at last visit, approximately 10 weeks later)
  Measures the number of meters the participant can walk in 6 minutes at a self-selected pace.
Functional outcome measure: Change from baseline in KOOS (Knee Injury and Osteoarthritis Outcome Score) to Post-Treatment | Baseline (measured at first visit) and post-treatment (measured at last visit, approximately 10 weeks later)
  The KOOS is a self-reported survey containing five subscales, each of which is considered separately (i.e. there is no "total" KOOS score). The investigators will use three of the KOOS subscales: Pain (Minimum Detectable Change [MDC] 13.4 points for people with KOA), Activities of Daily Living (MDC 15.4 points), and Quality of Life (MDC 21.1 points). Each subscale is measured on a 0-100 scale, with lower scores indicating worse symptoms / worse function.

CONTACTS AND LOCATIONS:
Overall Officials: Allyn Bove, DPT, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Only fully deidentified data will be made available to other researchers upon request and approval by the investigators and the relevant institutional review board.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available upon the conclusion of the study for up to seven years upon request.
Access Criteria: Requests for data sharing must be agreed to by the investigators and the relevant institutional review board.